CLINICAL TRIAL: NCT03213236
Title: OSA Homemonitoring
Acronym: OSA+
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancelled during overtaking maneuver
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S60319
Record Dates: First submitted 2017-06-27; First posted 2017-07-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OSA Homemonitoring (Experimental): Homemonitoring diagnostic system
  Interventions: Diagnostic Test: Homemonitoring diagnostic system

INTERVENTIONS:
Diagnostic Test: Homemonitoring diagnostic system — In addition to the standard full-night diagnostic polysomnography, patients will be evaluated during the same night with a "homemonitoring diagnostic system" that consists out of a pulse oximeter, accelerometer, smartphone for audio recording and a mattress that measures the ballistocardiogram.

SUMMARY:
Up to now, no studies are available where a comparison has been made between the accuracy of, on the one hand, the gold standard PSG and, on the other hand, a home monitoring sleep apnea-diagnostic system, consisting of a pulse oximeter, and accelerometer, a smartphone for snoring analysis, and a mattress for ballistocardiographic (BCG) recordings.

The purpose of this study is twofold. On the one hand, a comparison between the predictive performance of an automated home monitoring system and the gold standard PSG in sleep apnea diagnosis will be performed. The home monitoring system consists of a pulse oximeter, an accelerometer, a smartphone to record ambient sound, and a mattress to record the BCG signal. This system will be provided by KU Leuven and Equilli, two partners that work together with the Sleep Laboratory at UZ Leuven and the group STADIUS of the KU Leuven in the OSA+ project. The system performs automated signal processing and classification in order to determine the presence of sleep apnea events. On the other hand, this study aims to improve the phenotyping of patients suffering from sleep apnea. This task will be first developed using the classical PSG and later an evaluation will be performed on the less obtrusive system.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the sleep lab for a diagnostic polysomnography because of suspicion of sleep apnea will be considered to participate in the trial upon signature of the informed consent.

Exclusion Criteria:

* Patients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the homemonitoring system | 1 day
  Accuracy of the homemonitoring system of apnea/hypopnea index measurement (in comparison with gold standard) polysomnography)

SECONDARY OUTCOMES:
Cardiovascular risk prediction tool | 1 day
  The homemonitoring system will lead to new signals that could better predict cardiovascular risk in comparison with the apnea/hypopnea index of the polysomnography. This tool will be based on a new algorithm that will be developed based on the results.
Apnea/hypopnea index severity | 1 day
  Evaluation of agreement between patient categorisation into apnea severity categories obtained by the homemonitoring system and the diagnostic polysomnography scoring

CONTACTS AND LOCATIONS:
Overall Officials: Bertien Buyse, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No